CLINICAL TRIAL: NCT02846259
Title: The Clinical Benefit and Risk of Oral Aspirin for Patients Who Have Unruptured Intracranial Aneurysm Combined With Cerebral Ischemia
Brief Title: The Clinical Benefit and Risk of Oral Aspirin for Unruptured Intracranial Aneurysm Combined With Cerebral Ischemia
Acronym: CBROAUNACCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Beijing Chao Yang Hospital (Other); Beijing Friendship Hospital (Other); The Second Hospital of Hebei Medical University (Other); Tianjin Medical University General Hospital (Other); Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, principal, Beijing Tiantan Hospital
Other Study IDs: SKW2016-13-aspirin
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Intracranial Aneurysm; Cerebral Ischemia
Keywords: intracranial aneurysm; cerebral ischemia; aspirin
MeSH Terms: conditions — Intracranial Aneurysm; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The first purpose of this study is to find out the clinical benefit and risk of oral aspirin for unruptured intracranial aneurysm (small than 7mm) combined with cerebral ischemia in patients in the real world.

The second purpose of this study is to get the prediction model of aneurysm's rupture in patients who has unruptured intracranial aneurysm (small than 7mm) combined with cerebral ischemia , and find out who is suitable for oral aspirin.

DETAILED DESCRIPTION:
The investigators try to collect the information of the patients have unruptured intracranial aneurysm combined with cerebral ischemia when oral aspirin.The characteristics of this study are large sample, multi center and prospective.In the real world, more and more patients are checked out unruptured intracranial aneurysm combined with cerebral ischemia.The investigators can collect the information such as how they use aspirin (dose, frequency, duration of treatment), demographic information, past history, daily life habits, morphological characteristics of the aneurysm, how they use other antithrombotic drugs.The investigators will record whether the aneurysm ruptured and have hemorrhage, ischemic stroke, death, changes in the morphology of aneurysm, MRI permeability image index changes. Finally the investigators will get the clinical benefits and risks of using aspirin and build the prediction model of rupture and hemorrhage for aneurysm, find out who is suitable for oral aspirin.

ELIGIBILITY:
Inclusion Criteria:

1. has the diagnosis of unruptured intracranial aneurysm (using the CTA/DSA,smaller than 7mm)
2. has the history of TIA or any other diseases of cerebral ischemia
3. older than 18 years old
4. sign the informed consent

Exclusion Criteria:

1. has the history of intracranial aneurysm rupture hemorrhage or has more than one aneurysm untreated
2. has a family history of intracranial aneurysm
3. has AVM，MMD, intracranial tumor, hydrocephalus or intracranial hemorrhage
4. refuse to sign the informed consent
5. allergic to contrast medium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators chose the patiens from the Tiantan hospital and other hospitals that participated in this study.The patients will all have unruptured intracranial aneurysm with the history of cerebral ischemia.
Sampling Method: Non-Probability Sample
Enrollment: 2135 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Aneurysm rupture hemorrhage | 2 years during the follow-up period
  Aneurysm subarachnoid hemorrhage without trauma

SECONDARY OUTCOMES:
TIA | 2 years during the follow-up period
Aneurysm changing | 2 years during the follow-up period
  the aneurysm becomes bigger, its form changes, becomes two or more
dead | 2 years during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Yong Cao, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Weng J, Li H, Jiao Y, Fu W, Huo R, Yan Z, Xu H, Zhan J, Wang S, Du X, Cao Y, Zhao J. Atorvastatin and growth, rupture of small unruptured intracranial aneurysm: results of a prospective cohort study. Ther Adv Neurol Disord. 2021 Apr 9;14:1756286420987939. doi: 10.1177/1756286420987939. eCollection 2021. PMID 33953800
- [Derived] Weng JC, Wang J, Du X, Li H, Jiao YM, Fu WL, Huo R, Yan ZH, Xu HY, Wang S, Cao Y, Zhao JZ; Small Unruptured Aneurysms Study Group. Safety of Aspirin Use in Patients With Stroke and Small Unruptured Aneurysms. Neurology. 2021 Jan 5;96(1):e19-e29. doi: 10.1212/WNL.0000000000010997. Epub 2020 Oct 14. PMID 33055274
- [Derived] Weng JC, Wang J, Li H, Jiao YM, Fu WL, Huo R, Yan ZH, Xu HY, Zhan J, Wang S, Du X, Cao Y, Zhao JZ; Small Unruptured Aneurysms Study Group. Aspirin and Growth of Small Unruptured Intracranial Aneurysm: Results of a Prospective Cohort Study. Stroke. 2020 Oct;51(10):3045-3054. doi: 10.1161/STROKEAHA.120.029967. Epub 2020 Sep 3. PMID 32878566